CLINICAL TRIAL: NCT02794363
Title: Autologous Platelet Rich Plasma Intradermal Injections for Vulvar Lichen Sclerosus
Brief Title: Platelet Rich Plasma Injections for Vulvar Lichen Sclerosus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Vulvovaginal Disorders (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 604763-1
Record Dates: First submitted 2016-05-25; First posted 2016-06-09 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Lichen Sclerosus
MeSH Terms: conditions — Lichen Sclerosus et Atrophicus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autologous platelet rich plasma (Other): Autologous platelet rich plasma injection into vulvar skin. There are no placebo, sham, or active comparator arms
  Interventions: Biological: Autologous platelet rich plasma

INTERVENTIONS:
Biological: Autologous platelet rich plasma — 5cc of autologous platelet rich plasma derived from 50cc of whole blood will be injected into vulvar skin.

SUMMARY:
15 patients with biopsy proven active vulvar lichen sclerosus will be recruited by a clinic specializing in vulvar disorders. This study consists of a 2 week screening period and a 12-week treatment period. Participants will receive two separate treatments of autologous platelet rich plasma separated by 6 weeks. A repeat biopsy will be performed 6 weeks after the second autologous platelet rich plasma injection

DETAILED DESCRIPTION:
15 patients with biopsy proven active vulvar lichen sclerosus will be recruited by a clinic specializing in vulvar disorders. This study consists of a 2 week screening period. A 4mm vulvar punch biopsy will be obtained at the initiation of the screening period to confirm that the participant have active lichen sclerosus. 12 weeks after the biopsy, the participants will receive an injection of 5cc of autologous platelet rich plasma into the affected vulvar skin. Six weeks later, participants will receive an additional injection of 5cc of autologous platelet rich plasma. A repeat biopsy will be performed 6 weeks after the second autologous platelet rich plasma injection. The inflammation on both biopsy specimens will be determined by a dermatopathologist.

ELIGIBILITY:
Inclusion Criteria:

* Active lichen sclerosus
* no current treatment
* symptomatic 4/10 on visual analogue scale

Exclusion Criteria:

* history of vulvar carcinoma or VIN

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-05; Primary Completion 2016-01 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Decrease in inflammation on post treatment biopsies | 14 weeks
  Pathologist will grade inflammation on 0-4 scale of pre and post treatment biopsies

SECONDARY OUTCOMES:
Decrease in Pruritus | 14 weeks
  Participants will fill out a 10cm visual analogue scale that grade the amount of their pruritus (itching)
Investigator Global Assessment | 14 weeks
  The investigator will rate the severity of lichen sclerosus based on the amount of lichenification, fissures, and ulceration. This will be a 4 point scale.

IPD SHARING:
Plan to Share IPD: No